CLINICAL TRIAL: NCT05929482
Title: A Randomized Controlled Pilot Study to Examine the Impact of a Filmed Dramatized Story Intervention (Telenovela/Soap Opera) for HIV Prevention in Latinas.
Brief Title: Impact of a Telenovela/Soap Opera for HIV Prevention in Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0630; 1R34DA053887-01A1 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-07-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: HIV; Latinas; Primary Disease Prevention; Internet Based Intervention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: 2 arms, intervention and wait-listed control group. Participants in the intervention group will receive the 4 episodes of the Love infection intervention (one episode weekly) after the baseline assessment. Participants in the wait-listed control group will receive the intervention after completing the 6-month assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infección de Amor (Infectious Love) (Experimental): 71 Latinas will view four IA intervention episodes, one per week immediately after the baseline survey and orientation. Participants will receive an email to their preferred email address with a password to access to the episode on the IA's website: www.telenoveladeamor.com Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection). The one week time frame for each episode is needed to provide time to review and reflect about IA's content and modify HIV prevention behaviors. It will also allow Latinas to obtain information and support from the team and referral if needed. This time frame was effective to improve behaviors in previous studies.
  Interventions: Behavioral: Infección de Amor (Infectious Love)
- Wait-listed (Experimental): A wait-listed control group of 71 Latinas will receive IA in the same manner as the intervention group. Latinas will start watching the telenovela episodes 7 months after their baseline survey (after T3 survey). Latinas will be informed at recruitment of this group condition and the study randomization. During the waiting time, participants will be called on a monthly basis to encourage participation and refer to services if needed.
  Interventions: Behavioral: Infección de Amor (Infectious Love)

INTERVENTIONS:
Behavioral: Infección de Amor (Infectious Love) — Infectious Love is a filmed dramatized story (telenovela/soap opera) culturally tailored for US Latinas and delivered online.
  IA is a four-episode HIV prevention telenovela co-created with Latinas and a community-based participatory and interdisciplinary. Participants have one week window to watch the 10-minute episodes from their preferred device and location.

SUMMARY:
Latinas continue to be affected disproportionally by HIV in the United States (US). Often, Latinas are not aware of their HIV status. Also, their perception of low risk for HIV interferes with condom use, HIV testing and lack of awareness, access, and use of Pre-exposure Prophylaxis [PrEP]. About 60% of total HIV cases in NC occur among women of childbearing age, thus vulnerability to HIV is particularly acute among Latinas between ages 18 and 44 years old, an age group with the highest rate of new HIV infections in NC. These disparities indicate that HIV prevention among Latinas is urgent; therefore, the investigators propose an innovative intervention - a filmed dramatized story (telenovela/soap opera) Infección de Amor [IA] (Love Infection) - culturally tailored for Latinas in the US and delivered online. Infección de Amor was filmed and developed but has not been tested with the target audience. The proposed study will pilot test IA and move the intervention to online using a website that will allow individual access around the clock from any location and device, such as a smartphone, ensuring wide dissemination of the intervention in the future. This is a a two-year planning grant (R34) to prepare for an R01 efficacy trial. The aims are to: 1) Develop the intervention delivery website, conduct a website usability test, and test the feasibility and acceptability of the IA intervention (four telenovela episodes) with 10 Latinas, 2) Conduct a randomized controlled pilot study to examine change in HIV prevention behaviors (condom use; HIV testing; and PrEP awareness, access, and use) comparing 71 intervention and 71 control Latinas from baseline (Time 1 [T1], 0 months) to post-active intervention (Time 2 [T2], 1 month), and to six months follow-up, a period with no contact from the study staff (Time 3 [T3, 7 months]), and 3) Complete establishing the study infrastructure, expanding the multidisciplinary team, building the research partnerships with the community, finalize the protocol and training materials, refine recruitment and retention strategies, data collection and data management procedures, and obtain institutional review board approval in preparation for an R01 efficacy study. This study address the National Institute on Drug Abuse (NIDA) goal #4: increase NIDA research and programs' public impact. This is a novel intervention to advance HIV prevention for Latinas. This study implement a culturally durable and feasible intervention for Latinas.

DETAILED DESCRIPTION:
Aim 1. A total of 10 participants will be enrolled for aim 1 (Develop the intervention delivery website, conduct a website usability test, and test the feasibility and acceptability of the IA intervention (four telenovela episodes). This part of the study is not a randomized clinical trial. These participants will provide feedback about the usability of the intervention website. Usability testing will use approaches for recruitment, eligibility criteria, and retention protocols as planned for the Randomized Clinical Trial (RCT) pilot. As with the RCT pilot, women recruited for the usability testing will sign a consent form before participating. During usability testing, Latinas will receive: (a) username and password information, and a link to the website, (b) an online orientation to the website, (c) all the telenovela website sections including IA telenovela episodes, study measures, and access to referral information), (d) reminders about their participation using an automated notification system on the website. Latinas will receive a small incentive to compensate them for their time. After participants complete the usability test (approximately one month after the online orientation), they will complete the 10-item System Usability Scale that measures digital intervention usability. Items are scored on a 5-item Likert scale (strongly disagree to strongly agree). Based on Latinas' responses, changes to the IA website or study protocols will be made before the RCT pilot. If this is the case, an amendment to the protocols will be submitted later. Details of the Usability Testing of IA are described below.

Randomized Clinical Trial (Aim 2). A total of 142 participants will be enrolled to examine change in HIV prevention behaviors (condom use; HIV testing; and Pre-exposure Prophylaxis [PrEP] awareness, access, and use) comparing 71 intervention and 71 control Latinas from baseline (Time 1 [T1], 0 months) to post-active intervention (Time 2 [T2], 1 month), and to six months follow-up, a period with no contact from the study staff (Time 3 [T3, 7 months]) Inclusion criteria are: Latinas ages 18-44 years who report sexual activity with a man in the last 6 months, have internet access from any device, and reside in NC. The research team is bilingual and will be able to assist women if they have questions about the study. Study procedures will be conducted in English and/or Spanish according to participant's preference. Recruitment and screening will be led by a bilingual (English and Spanish) study personnel. Participants will be asked their preferred language at the time of recruitment. All study materials, including information and consent forms, questionnaires, and recruitment ads, will be translated and available in Spanish. Any direct interaction with non-English-speaking participants will be available in Spanish.

The study is targeting a minority population in the United States, and special efforts will be made to make the study attractive for them, such as offering recruitment flyers, measures and consent forms in Spanish and English; referral health centers that are accessible for, if needed; and study team personnel who are culturally sensitive to the Latinas' culture.

Infección de Amor website. The website will provide: a) access to the four intervention episodes 24/7 from any location or type of device (e.g., cellphone, laptop) since it will be mobile optimized (all the episodes are password protected); b) questionnaires for data collection deployed via Qualtrics; c) a contact section in case participants have technical problems or need to contact the research team; and d) a section with community resources, services, and referrals. Secure and private servers and communication channels will be used such as OneDrive/Microsoft teams to store and to exchange information.

The intervention website will be accessible to study participants in English and Spanish. The intervention participants will access telenovela episodes, available in Spanish or English, at their preferred time and place using a website accessible through any device since it will be mobile optimized. A new episode of IA will be available each week. Women will be instructed to watch an episode as many times as they want during the week, but they need to answer a post episode-viewing survey after viewing it the first time. Also, they will be able to pause or stop the episodes at any time if they need to take a break or stop watching for any reason. Women will be advised to watch the episodes alone. Prior episodes will remain available after a new episode is released. Each episode has an opening that introduces the characters and then the content of the telenovela.

Participants will receive reminders about completion of the surveys. In addition, up to three reminders (e.g., phone, email) will be sent each week to participants who have not accessed an episode in a specific window period and completed the post episode survey or if the participant has not access to the website in one week. If a woman does not complete the episode in one week or does not access the website in one week, the research team will contact the participant (e.g., emails, calls, or text messages) to her preferred email or phone. The research team will discuss with her any impediments to her participation, how to watch the missed episode, and resume with the following episodes. Women will be able to pause or stop the episodes at any time if they need it. Prior episodes will remain available after a new episode is released if women would like to review them.

Recruitment and enrollment. The investigators will enroll 60-64 Latinas per quarter (5-6 per week). If needed, enrollment timeline can be extended and advice from health departments and Dr. Barrington will be requested if there are issues enrolling participants. A standardized eligibility form will be used to assess if Latinas meet inclusion criteria (e.g., age, internet access) that will be available in Qualtrics.

Baseline survey. If potential participants meet the inclusion criteria, they will be asked to attend to a one hour-meeting with a member of the research team to sign the informed consent, complete a baseline survey and receive an orientation about the use of the telenovela website. After participants complete the survey, they will be randomized by a member of the research team to the intervention or control group. The research team will randomize participants to the intervention and control groups by a computer-generated randomization table, using blocking of participants to ensure a balance between groups in relation to participant's characteristics (e.g., presence of substance abuse [SA], intimate partner violence [IPV], or depression), and participants will be informed of their group assignment by phone. The research team member will explain the following activities they have to complete according to the group they will be assigned. If they are randomized to the control group, the orientation to the website will be delayed until they complete the 7-month post baseline survey. The survey will be available in Qualtrics and only the members of the research team will have access to the survey.

Intervention group: 71 Latinas will view four Infección de Amor (IA, Love Infection) intervention episodes, one per week. Participants will receive an email to their preferred email address with a password to access to the episode on the IA's website.

Each 10-minute episode can be watched more than once during the week and presents a situation with notable HIV risk and ways the characters avoided risk (e.g., condom use) or confronted consequences of poor practices (e.g., HIV infection). The one-week time frame for each episode is needed to provide time to review and reflect about IA's content and modify HIV prevention behaviors. It will also allow Latinas to obtain information and support from the team and referral if needed. This time frame was effective to improve behaviors in previous studies.

After each episode, participants will complete a survey (on their own) on Qualtrics. This post episode survey includes questions about the mechanisms of action of the telenovela (self-efficacy, narrative engagement, and emotional elicitation).

Control group: A wait-listed control group of 71 Latinas will receive IA in the same manner as the intervention group after completing T3 data collection. Latinas will be informed at recruitment of this group condition and the study randomization. During the waiting time, participants will be called on a monthly basis to encourage participation and refer to services if needed.

Follow-up surveys. Participants will answer a (one-month after baseline) survey, and complete another survey (on their own) 7 months after baseline. Participants will complete these surveys (1-month and 7-months after baseline) on their own. Participants can request help to complete these surveys (online using zoom or face to face if needed). Zoom meetings will not be recorded if the surveys are conducted using zoom.

Procedures for Minority Retention and Potential Challenges. For each video episode, participants will have a one-week window to view and will receive reminders using an automated notification system from Qualtrics when the end of the viewing-window is approaching. The website will track if participants watch the whole episode. Information about HIV prevention will be provided at the end of each episode and a link to the technical support and referrals sections if needed. Other retention strategies will include: 1) updating contact information frequently; 2) requesting contact information of at least two friends or relatives; 3) contacting the woman by email or cell phone (permission in the informed consent will be requested for contacting them); 4) providing compensation for their time, internet use, and transportation; and 5) automated notification system messages for special occasions (e.g., holidays). The researchers will be flexible in scheduling enrollment and data collection appointments. Attrition will be monitored in both conditions. Potential issues with Latinas and community centers will be discussed, and if needed, a community advisory board of three Latinas of the same age as those participating in the study to ask for their advice will be established. Participants will receive a compensation for their participation in the study.

Fidelity of the Intervention. The NIH five-category treatment Fidelity Framework will be used. For study design, the theoretical model was articulated; Latinas in both intervention and wait-listed control groups will receive the same telenovela intervention at different times. Also an optimal protocol will be created to ensure that the intervention is fully operationalized.

Variables and their measurement. The measures will be available in Spanish and English; in previous studies with Latinas, they demonstrated excellent reliability and validity and are written at a 4th-grade reading level. Measures available in Spanish and English that are part of the PhenX toolkit recommended by the NIDA were added, including: a) sociodemographic information (e.g., income, housing situation); b) questionnaires at each timepoint assessing HIV behavioral outcomes and moderators of HIV prevention behaviors; c) post-IA episode surveys measuring the mechanisms of action.

All study personnel will be adult, bilingual, and will receive training in human subjects and a 3-5 day training about study procedures and their specific functions in the study (e.g., website access, use of Qualtrics, and Microsoft excel).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as a Latina
* Assigned female gender at birth
* Fluent in English or Spanish
* Between 18 and 44 years old
* Report sexual activity with a man in the last 6 months
* Have internet access from any device
* Reside in NC

Exclusion Criteria:

* Unwilling to be part of the study
* Do not read, speak, or understand Spanish or English
* Do not have access to internet
* HIV positive

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study includes female Latinas between 18 and 44 years old. Older women (>44 years old) and younger children/adolescents (<18) are excluded.
Enrollment: 95 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Condom Use from Baseline to Month 1 | baseline up to 1 month
  Changes in condom use will be measured as the number of sexual episodes (oral, vaginal, or anal intercourse) in which condoms were used with a male partner in the last month.
Change in Condom Use from Baseline to Month 7 | baseline up to 7 months
  Changes in condom use will be measured as the number of sexual episodes (oral, vaginal, or anal intercourse) in which condoms were used with a male partner in the last month.
Changes in Pre-exposure Prophylaxis [PrEP] Awareness from Baseline to Month 1 | baseline up to 1 month
  Changes in PrEP awareness will be measured as the number of participants who self-report whether they know about PrEP medication (dichotomous question: yes/no)
Changes in Pre-exposure Prophylaxis [PrEP] Awareness from Baseline to Month 7 | baseline up to 7 months
  Changes in PrEP awareness will be measured as the number of participants who self-report whether they know about PrEP medication (dichotomous question: yes/no)
Changes in Pre-exposure Prophylaxis [PrEP] Access from Baseline to Month 1 | baseline to 1 month
  Changes in PrEP access will be measured as the number of participants who report that they have access to PrEP (dichotomous question: yes/no)
Changes in Pre-exposure Prophylaxis [PrEP] Access from Baseline to Month 7 | baseline to 7 months
  Changes in PrEP access will be measured as the number of participants who report that they have access to PrEP (dichotomous question: yes/no)
Changes in Pre-exposure Prophylaxis [PrEP] Use from Baseline to Month 1 | baseline to 1 month
  Changes in PrEP use will be measured as the number of participants who self-report whether they use PrEP medication (dichotomous question: yes/no)
Changes in Pre-exposure Prophylaxis [PrEP] Use from Baseline to Month 7 | baseline up to 7 months
  Changes in PrEP use will be measured as the number of participants who self-report whether they use PrEP medication (dichotomous question: yes/no).
Change in HIV Testing from Baseline to Month 1 | baseline up to 1 month
  Changes in HIV testing will be measured as the number of participants who reported to have been tested for HIV in the last month.
Change in HIV Testing from Baseline to Month 7 | baseline up to 7 months
  Changes in HIV testing will be measured as the number of participants who reported to have been tested for HIV in the last month.
Change in HIV Test Perception from Baseline to Month 1 | baseline up to 1 month
  Changes in HIV testing perception will be measured with the willingness to take an HIV test measure scale. Scores range from 9-45. A higher score represents a higher willingness to take an HIV test.
Change in HIV Test Perception from Baseline to Month 7 | baseline up to 7 months
  Changes in HIV testing perception will be measured with the willingness to take an HIV test measure scale. Scores range from 9-45. A higher score represents a higher willingness to take an HIV test.

SECONDARY OUTCOMES:
Number of Participants who Complete all the Intervention Content | 40-minute
  The online website will track the number of participants who complete of all intervention content (40-minute of the telenovela episode)
Number of Participants Who are Retained Through all Assessments | baseline up to 7 months
  The number of participants who completed all assessments divided by the number of enrolled participants
Change in Emotional Response | Changes in emotional Response (ER) will be measured with the International Positive and Negative Affect Schedule Short Form (IPANAS-SF). Scores range from 10-50. Higher scores indicate the tendency to experience a positive and negative mood.
  Changes in emotional Response (ER) will be measured with the International Positive and Negative Affect Schedule Short Form (IPANAS-SF). Scores range from 10-50. Higher scores indicate the tendency to experience a positive and negative mood.
Change in Narrative Engagement | week 1 to week 4
  Changes in narrative engagement (NE) will be measured with the Perception of Narrative Performance Scale, which measures three dimensions of engagement: interest, realism, and identification. Scores range from 9-36. A higher score indicates a higher level of engagement.
Change in Self-Efficacy for Condom Use | week 1 to week 4
  Changes in Self-Efficacy for condom use will be measured using the HIV self-efficacy for condom use survey. Scores range from 7-28. A higher score indicates a higher level of self-efficacy for condom use.
Emotional response, narrative engagement, and self efficacy as predictors of condom use | one month to 7 months post baseline
  The effects of emotional response (ER), Narrative engagement (NE) and Self-efficacy (SE) on condom use will be estimated. ER, NE and SE will be measured using the scales reported on outcomes 15-17 and condom use will be measured as described in outcome 1. A lineal regression model including group assignment (intervention or control), ER, NE and SE as predictors of condom use will be conducted. The estimated regression coefficients (beta) of each independent variable will be reported. Higher estimated regression coefficients represent higher effects of these variables on condom use.
Emotional response, narrative engagement, and self efficacy as predictors of HIV testing | one month to 7 months post baseline
  The effects of emotional response (ER), Narrative engagement (NE) and Self-efficacy (SE) on HIV testing will be estimated. ER, NE and SE will be measured using the scales reported on outcomes 15-17 and HIV testing will be measured as described in outcome 9. A logistic regression model will be conducted including group assignment (intervention or control), ER, NE and SE as predictors of HIV testing. The estimated odd ratios of each predictor will be reported. Odds ratio greater than 1 will indicate higher occurrence of HIV testing given exposure to the predictors.
Emotional response, narrative engagement, and self efficacy as predictors of PrEP awareness | one month to 7 months post baseline
  The effects of emotional response (ER), Narrative engagement (NE) and Self-efficacy (SE) on PrEP awareness will be estimated. ER, NE and SE will be measured using the scales reported on outcomes 15-17 and PrEP awareness will be measured as described in outcome 3. A logistic regression model will be conducted including group assignment (intervention or control), ER, NE and SE as predictors of PrEP awareness. The estimated odd ratios of each predictor will be reported. Odds ratio greater than 1 will indicate higher occurrence of PrEP awareness given exposure to the predictors.
Change in Substance Abuse from Baseline to Month 7 | baseline up to 7 months
  Changes in substance abuse will be measured with the Substance abuse behaviors scale. Scores range from 6-36. A higher score represents a higher use of substances.
Change in Intimate Partner Violence (IPV) | baseline up to 7 months
  Changes in IPV will be measured using the revised Conflict Tactics Scale to measure women's self-reported IPV in the previous 3 months (e.g., your partner insulted you). Scores range from 24-72 points. A higher score indicates higher levels of IPV.
Change in Depression | baseline up to 7 months
  Changes in depression will be measured with the Patient Health screening in primary care and other health settings. Scores range from 5-27. A higher score indicates more depressive symptoms.
Substance abuse, intimate partner violence, and depression as predictors of condom use | baseline up to 7 months
  Substance abuse (SA), intimate partner violence (IPV) and depression measured with the scales described in outcome 21-23 will be tested as predictors of condom use (measured as described outcome 1). A linear regression model will be conducted. The estimated regression coefficients (beta) of each predictor will be reported. Higher coefficients indicate a stronger effect of these variables on condom use.
Substance abuse, intimate partner violence, and depression as predictors of HIV testing | baseline up to 7 months
  Substance abuse (SA), intimate partner violence (IPV) and depression measured with the scales described in outcome 21-23 will be tested as predictors of HIV testing (measured as described outcome 9). A logistic regression model will be conducted. The estimated odds ratio of each independent variable will be reported. Odds ratio greater than 1 will indicate higher occurrence of HIV testing given exposure to the predictors.
Substance abuse, intimate partner violence, and depression as predictors of PrEP awareness | baseline up to 7 months
  Substance abuse (SA), intimate partner violence (IPV) and depression measured with the scales described in outcome 21-23 will be tested as predictors of PrEP awareness (measured as described outcome 3). A logistic regression model will be conducted. The estimated odds ratio of each predictor will be reported. Odds ratio greater than 1 will indicate higher occurrence of PrEP awareness given exposure to the predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia A Villegas Rodriguez, PhD, Principal Investigator — University of North Carolina at Chapel Hill School of Nursing
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and continuing for 36 months following publication
Access Criteria: Borrower has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.
URL: https://www.telenoveladeamor.com/

REFERENCES:
- [Background] Levison JH, Bogart LM, Khan IF, Mejia D, Amaro H, Alegria M, Safren S. "Where It Falls Apart": Barriers to Retention in HIV Care in Latino Immigrants and Migrants. AIDS Patient Care STDS. 2017 Sep;31(9):394-405. doi: 10.1089/apc.2017.0084. PMID 28891715
- [Background] Cianelli R, Ferrer L, McElmurry BJ. HIV prevention and low-income Chilean women: machismo, marianismo and HIV misconceptions. Cult Health Sex. 2008 Apr;10(3):297-306. doi: 10.1080/13691050701861439. PMID 18432428
- [Background] Villar-Loubet OM, Vamos S, Jones DL, Lopez E, Weiss SM. A Cultural Perspective on Sexual Health: HIV Positive and Negative Monolingual Hispanic Women in South Florida. Hisp Health Care Int. 2011 Jun 1;9(2):82-90. doi: 10.1891/1540-4153.9.2.82. PMID 24994949
- [Background] Cianelli R, Villegas N. Social Determinants of Health for HIV Among Hispanic Women. Hisp Health Care Int. 2016 Mar;14(1):4-9. doi: 10.1177/1540415316629672. No abstract available. PMID 27257185
- [Background] Sanchez M, Rojas P, Li T, Ravelo G, Cyrus E, Wang W, Kanamori M, Peragallo NP, De La Rosa MR. Evaluating a Culturally Tailored HIV Risk Reduction Intervention Among Latina Immigrants in the Farmworker Community. World Med Health Policy. 2016 Sep;8(3):245-262. doi: 10.1002/wmh3.193. Epub 2016 Sep 17. PMID 29034116
- [Background] Torrone EA, Wright J, Leone PA, Hightow-Weidman LB. Pregnancy and HIV infection in young women in North Carolina. Public Health Rep. 2010 Jan-Feb;125(1):96-102. doi: 10.1177/003335491012500113. PMID 20402201
- [Background] Paz K, Massey KP. Health Disparity among Latina Women: Comparison with Non-Latina Women. Clin Med Insights Womens Health. 2016 Jul 20;9(Suppl 1):71-4. doi: 10.4137/CMWH.S38488. eCollection 2016. PMID 27478393
- [Background] Garcia J, Perez-Brumer AG, Cabello R, Clark JL. "And Then Break the Cliche": Understanding and Addressing HIV Vulnerability Through Development of an HIV Prevention Telenovela with Men Who Have Sex with Men and Transwomen in Lima, Peru. Arch Sex Behav. 2018 Oct;47(7):1995-2005. doi: 10.1007/s10508-017-1119-x. Epub 2018 Feb 20. PMID 29464455
- [Background] Zou B, Jin B, Koch GG, Zhou H, Borst SE, Menon S, Shuster JJ. On model selections for repeated measurement data in clinical studies. Stat Med. 2015 May 10;34(10):1621-33. doi: 10.1002/sim.6414. Epub 2015 Jan 23. PMID 25645442
- [Background] Center for Disease Control and Prevention (CDC). Women and HIV: Where we are going. https://www.hiv.gov/blog/cdc-women-and-hiv-where-we-are-going. Updated 2019
- [Background] Center for Disease Control and Prevention (CDC). HIV among women. https://www.cdc.gov/hiv/group/gender/women/index.html. Updated 2020
- [Background] MedPage Today. PrEP use among heterosexual women. https://www.medpagetoday.com/resource-centers/contemporary-hiv-prevention/prep-use-among-heterosexual-women/1593. Updated 2020.
- [Background] Alvidrez J, Castille D, Laude-Sharp M, Rosario A, Tabor D. The National Institute on Minority Health and Health Disparities Research Framework. Am J Public Health. 2019 Jan;109(S1):S16-S20. doi: 10.2105/AJPH.2018.304883. PMID 30699025
- [Background] Wingood GM, DiClemente RJ, Villamizar K, Er DL, DeVarona M, Taveras J, Painter TM, Lang DL, Hardin JW, Ullah E, Stallworth J, Purcell DW, Jean R. Efficacy of a health educator-delivered HIV prevention intervention for Latina women: a randomized controlled trial. Am J Public Health. 2011 Dec;101(12):2245-52. doi: 10.2105/AJPH.2011.300340. Epub 2011 Oct 20. PMID 22021297
- [Result] Larkey LK, Hecht ML, Miller K, Alatorre C. Hispanic cultural norms for health-seeking behaviors in the face of symptoms. Health Educ Behav. 2001 Feb;28(1):65-80. doi: 10.1177/109019810102800107. PMID 11213143
- [Result] Miller-Day M, Hecht ML. Narrative means to preventative ends: a narrative engagement framework for designing prevention interventions. Health Commun. 2013;28(7):657-70. doi: 10.1080/10410236.2012.762861. Epub 2013 Aug 27. PMID 23980613
- [Result] Nabi RL. Emotional flow in persuasive health messages. Health Commun. 2015;30(2):114-24. doi: 10.1080/10410236.2014.974129. PMID 25470436
- [Result] Nabi RL. Laughing in the Face of Fear (of Disease Detection): Using Humor to Promote Cancer Self-Examination Behavior. Health Commun. 2016 Jul;31(7):873-83. doi: 10.1080/10410236.2014.1000479. Epub 2015 Dec 11. PMID 26652312
- [Result] Geter Fugerson A, Sutton MY, Hubbard McCree D. Social and Structural Determinants of HIV Treatment and Care Among Hispanic Women and Latinas Living with HIV Infection in the United States: A Qualitative Review: 2008-2018. Health Equity. 2019 Nov 4;3(1):581-587. doi: 10.1089/heq.2019.0039. eCollection 2019. PMID 31701083
- [Result] Peragallo N, Deforge B, O'Campo P, Lee SM, Kim YJ, Cianelli R, Ferrer L. A randomized clinical trial of an HIV-risk-reduction intervention among low-income Latina women. Nurs Res. 2005 Mar-Apr;54(2):108-18. doi: 10.1097/00006199-200503000-00005. PMID 15778652
- [Result] Peragallo Montano N, Cianelli R, Villegas N, Gonzalez-Guarda R, Williams WO, de Tantillo L. Evaluating a Culturally Tailored HIV Risk Reduction Intervention Among Hispanic Women Delivered in a Real-World Setting by Community Agency Personnel. Am J Health Promot. 2019 May;33(4):566-575. doi: 10.1177/0890117118807716. Epub 2018 Oct 24. PMID 30354190
- [Result] Villegas N, Santisteban D, Cianelli R, Ferrer L, Ambrosia T, Peragallo N, Lara L. The development, feasibility and acceptability of an Internet-based STI-HIV prevention intervention for young Chilean women. Int Nurs Rev. 2014 Mar;61(1):55-63. doi: 10.1111/inr.12080. PMID 24512261
- [Result] Villegas N, Santisteban D, Cianelli R, Ferrer L, Ambrosia T, Peragallo N, Lara L. Pilot testing an internet-based STI and HIV prevention intervention with Chilean women. J Nurs Scholarsh. 2015 Mar;47(2):106-16. doi: 10.1111/jnu.12114. Epub 2014 Nov 19. PMID 25410132
- [Result] Cianelli R, Ferrer L, Norr KF, Miner S, Irarrazabal L, Bernales M, Peragallo N, Levy J, Norr JL, McElmurry B. Mano a Mano-Mujer: an effective HIV prevention intervention for Chilean women. Health Care Women Int. 2012;33(4):321-41. doi: 10.1080/07399332.2012.655388. PMID 22420675
- [Result] Sikkema KJ, Heckman TG, Kelly JA, Anderson ES, Winett RA, Solomon LJ, Wagstaff DA, Roffman RA, Perry MJ, Cargill V, Crumble DA, Fuqua RW, Norman AD, Mercer MB. HIV risk behaviors among women living in low-income, inner-city housing developments. Am J Public Health. 1996 Aug;86(8):1123-8. doi: 10.2105/ajph.86.8_pt_1.1123. PMID 8712272
- [Result] Heckman T, Kelly J, Sikkema K, et al. HIV risk characteristics of young adult, adult, and older adult women who live in inner-city housing developments: Implications for prevention. J Women's Health Gend Based Med. 1995;4(4):397-406.
- [Result] Garcia M, Harris AL. PrEP awareness and decision-making for Latino MSM in San Antonio, Texas. PLoS One. 2017 Sep 27;12(9):e0184014. doi: 10.1371/journal.pone.0184014. eCollection 2017. PMID 28953905
- [Result] Cianelli R, Villlegas N, De Oliveira G, Hires K, Gattamorta K, Ferrer L, Peragallo N. Predictors of HIV enacted stigma among Chilean women. J Clin Nurs. 2015 Sep;24(17-18):2392-401. doi: 10.1111/jocn.12792. Epub 2015 Feb 19. PMID 25693422
- [Result] Catania J. Dyadic sexual communication scale: Handbook of sexuality related measures. 1986.
- [Result] Catania JA, Kegeles SM, Coates TJ. Towards an understanding of risk behavior: an AIDS risk reduction model (ARRM). Health Educ Q. 1990 Spring;17(1):53-72. doi: 10.1177/109019819001700107. PMID 2318652
- [Result] Kelly JA, Murphy DA, Washington CD, Wilson TS, Koob JJ, Davis DR, Ledezma G, Davantes B. The effects of HIV/AIDS intervention groups for high-risk women in urban clinics. Am J Public Health. 1994 Dec;84(12):1918-22. doi: 10.2105/ajph.84.12.1918. PMID 7998630
- [Result] Straus MA, Douglas EM. A short form of the Revised Conflict Tactics Scales, and typologies for severity and mutuality. Violence Vict. 2004 Oct;19(5):507-20. doi: 10.1891/vivi.19.5.507.63686. PMID 15844722
- [Result] Radloff LS. The CES-D scale: A self report depression scale for research in the general population. Appl Psychol Meas. 1977;1:385-401
- [Result] Card J, Solomon J, Berman J, eds. Tools for building culturally competent HIV prevention programs. New York: Springer Publishing Company; 2008.
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Lelutiu-Weinberger C, Golub SA. Enhancing PrEP Access for Black and Latino Men Who Have Sex With Men. J Acquir Immune Defic Syndr. 2016 Dec 15;73(5):547-555. doi: 10.1097/QAI.0000000000001140. PMID 27454250
- [Result] Bauermeister JA, Meanley S, Pingel E, Soler JH, Harper GW. PrEP awareness and perceived barriers among single young men who have sex with men. Curr HIV Res. 2013 Oct;11(7):520-7. doi: 10.2174/1570162x12666140129100411. PMID 24476355
- [Result] Walsh JL. Applying the Information-Motivation-Behavioral Skills Model to Understand PrEP Intentions and Use Among Men Who Have Sex with Men. AIDS Behav. 2019 Jul;23(7):1904-1916. doi: 10.1007/s10461-018-2371-3. PMID 30554396
- [Result] Blackstock OJ, Patel VV, Felsen U, Park C, Jain S. Pre-exposure prophylaxis prescribing and retention in care among heterosexual women at a community-based comprehensive sexual health clinic. AIDS Care. 2017 Jul;29(7):866-869. doi: 10.1080/09540121.2017.1286287. Epub 2017 Feb 1. PMID 28147704
- [Result] De Oliveira G, Cianelli R, Gattamorta K, Kowalski N, Peragallo N. Social Determinants of Depression Among Hispanic Women. J Am Psychiatr Nurses Assoc. 2017 Jan/Feb;23(1):28-36. doi: 10.1177/1078390316669230. Epub 2016 Sep 19. PMID 27624770

DOCUMENTS (1):
  • Informed Consent Form (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT05929482/ICF_000.pdf